CLINICAL TRIAL: NCT00479674
Title: A Phase II Study of Abraxane®, Carboplatin and Bevacizumab in "Triple Negative" (Demonstrating No Expression for Estrogen, Progesterone, or Her2 Receptors) Metastatic Breast Cancer
Brief Title: Phase II Study With Abraxane, Bevacizumab and Carboplatin in Triple Negative Metastatic Breast Cancer
Acronym: ABC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014837; AVF3962s
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer; Advanced Breast Cancer; Hormone Receptor AND Her2/neu Negative; Triple Negative; Triple Negative Breast Cancer; Stage IV or Inoperable Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Taxes; Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abraxane, Carboplatin, Bevacizumab (Experimental): Abraxane 100 mg/m2 IV over 30 min days 1,8,15.; Carboplatin AUC=2 IV over 15 min days 1,8,15., Bevacizumab 10 mg/kg IV days 1,15
  Interventions: Drug: Abraxane; Drug: Bevacizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Abraxane — 100 mg/m2 IV over 30 min days 1,8,15. Cycles Repeated Every 28 days until documented evidence of disease progression by RECIST criteria, intolerable toxicity, or death..
  Other Names: nanoparticle albumin-bound paclitaxel
Drug: Bevacizumab — 10 mg/kg IV days 1,15 Cycles Repeated Every 28 days until documented evidence of disease progression by RECIST criteria,intolerable toxicity, or death.
  Other Names: Avastin
Drug: Carboplatin — area under curve (AUC)=2 IV over 15 min days 1,8,15. Cycles Repeated Every 28 days until documented evidence of disease progression by RECIST criteria, intolerable toxicity, or death.

SUMMARY:
Taxanes (such as paclitaxel) are highly active to treat breast cancer. Abraxane® (nanoparticle albumin-bound paclitaxel) compared to standard paclitaxel improves efficacy and tolerability. When combined with a taxane, platinum agents improve response in metastatic breast cancer, with carboplatin conferring less toxicity than cisplatin. Monoclonal antibodies including bevacizumab target vascular endothelial growth factor (VEGF) to reduce angiogenesis. We hypothesize that the previously-untested combination of weekly Abraxane® and carboplatin plus biweekly bevacizumab will lengthen time to progression without producing intolerable toxicity.

DETAILED DESCRIPTION:
Anthracycline-based chemotherapy is widely used as adjuvant treatment for breast cancer. In addition to the challenge posed by anthracycline-induced cardiotoxicity, there are issues surrounding previous treatment with anthracyclines which limit its utility in the metastatic disease setting. Many patients with advanced disease will have had prior anthracycline-based adjuvant therapy, may have reached a maximum cumulative lifetime dose, or developed refractory disease, creating an obvious need for non-anthracycline treatment strategies.3 Platinum- and taxane-based chemotherapies as first-line therapy for metastatic breast cancer have demonstrated significant activity, producing single-agent response rates > 50%; in combination these rates increased to > 60% in both previously untreated and in patients who previously received anthracyclines.3 However, overall survival has remained relatively unchanged.4 As there is currently no standard of care for patients with metastatic breast cancer, various physical and psychological factors must be considered when evaluating chemotherapy treatment options, including the patient's tumor biology and growth rate, presence and extent of metastases, history of prior treatment and response, sensitivity and tolerance to therapy, and quality of life.2 Strategies to develop combination, higher dose, or sequential regimens using these active agents, while improving response rates and/or time to progression, may produce increased toxicity without increased survival.2 Because metastatic breast cancer remains essentially incurable using cytotoxic therapy alone, the study of targeted biologics offers new opportunities to enhance drug delivery via their ability to regulate specific receptors that are associated with clinically aggressive disease processes.

ELIGIBILITY:
Inclusion Criteria:

* Tissue block containing tumor to confirm metastatic breast cancer is required;
* Measurable disease according to RECIST criteria
* "Triple negative" disease defined as tumor demonstrating no expression for estrogen, progesterone or human epidermal growth factor receptor 2(HER2)receptors. "No expression" is categorized as ≤ 10% of cells staining or Allred ≤ 2;
* Aged 18 years or older;
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of 0 or 1; life expectancy ≥ 3 months;
* Patients may have received 0 - 1 prior therapies (except taxanes in the metastatic setting). An interval of at least 1 week must have elapsed since prior chemotherapy or hormonal therapy for metastatic disease; at least 6 months must have elapsed since prior adjuvant therapy;
* ≥ 2 weeks between surgery and study enrollment (≥ 4 weeks between major surgery (defined as open abdominal/thoracic/cardiac) and study enrollment;
* Laboratory tests performed within 14 days of study entry:

  * Granulocytes ≥ 1,500/µL;
  * Platelets ≥ 100,000/µL;
  * Hemoglobin ≥ 9 gm/dL;
  * Total bilirubin ≤ institutional upper limit of normal (ULN);
  * Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 5 times ULN;

    * Alkaline phosphatase ≤ 2.5 times ULN;
  * Estimated creatinine clearance ≥ 60 mL/min.
* left ventricular ejection fraction (LVEF)≥ 50% by multigated acquisition (MUGA)/Echocardiogram;
* Informed consent to receive protocol treatment, to provide biologic specimens, and to complete neurotoxicity questionnaires;
* Cognitive and communication skills to comply with study and/or follow-up procedures;
* No reproductive potential:

  * If pre-menopausal: Negative serum pregnancy test and patient agreement to use adequate contraceptive method (abstinence, intrauterine device, barrier device with spermicide or surgical sterilization) during and for 3 months after completion of treatment.
  * If post-menopausal: Amenorrhea for ≥ 12 months.

Exclusion Criteria:

* Pregnant or breast feeding;
* Prior treatment with Abraxane®, carboplatin or bevacizumab, or any taxane for metastatic breast cancer;
* Known hypersensitivity to any component of any study drug;
* Active infection;
* Current neuropathy ≥ grade 2;
* central nervous system (CNS) metastases as determined by head CT with contrast;
* History of bleeding within the past 6 months or active bleeding disorder;
* Serious non-healing wound, ulcer or bone fracture;
* Uncontrolled congestive heart failure (CHF), or history of myocardial infarction(MI), unstable angina, stroke, or transient ischemia within previous 6 months;
* Inadequately controlled hypertension (defined as systolic blood pressure < 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications; prior history of hypertensive crisis or hypertensive encephalopathy;
* Proteinuria (defined as urine protein: creatinine (UPC) ratio ≥ 1.0 or urine dipstick ≥ 2+.
* Significant vascular disease (aortic aneurysm, aortic dissection) or symptomatic peripheral vascular disease;
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within previous 6 months;
* Uncontrolled serious contraindicated medical condition or psychiatric illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Blackwell, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Presbyterian Health Care, Charlotte, North Carolina
  - Northeast Oncology Associates, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Forsyth Regional Cancer Center, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Jasim SA, Farber IM, Noraldeen SAM, Bansal P, Alsaab HO, Abdullaev B, Alkhafaji AT, Alawadi AH, Hamzah HF, Mohammed BA. Incorporation of immunotherapies and nanomedicine to better normalize angiogenesis-based cancer treatment. Microvasc Res. 2024 Jul;154:104691. doi: 10.1016/j.mvr.2024.104691. Epub 2024 May 3. PMID 38703993
- See also: Nab- Paclitaxel/Bevacizumab/Carboplatin chemotherapy in the first line triple negative metastatic breast cancer — http://dx.doi.org/10.1016/j.clbc.2013.08.003

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abraxane, Carboplatin, Bevacizumab
Started | 41
Completed | 0
Not Completed | 41
Not completed — Adverse Event | 18
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 14
Not completed — none provided | 3

BASELINE CHARACTERISTICS:
Arm/Group | Abraxane, Carboplatin, Bevacizumab
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 25
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Best Clinical Response Expressed as Percentage of Participants Treated With Combination Regimen of Weekly Abraxane® and Carboplatin Plus Biweekly Bevacizumab to Treat Women With Stage IV or Inoperable Stage III "Triple Negative" Metastatic Breast Cancer.
Description: Best clinical response is based on RECIST criteria, the proportion in each response category along with the exact binomial confidence intervals are estimated. Toxicity summaries are also provided.
Time Frame: 5 years
Population: 2 subjects withdrew and were not assessed for response
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abraxane, Carboplatin, Bevacizumab
Number analyzed (Participants) | 39
percentage of participants
  Complete Response | 18 [8 to 34]
  Partial Response | 69 [52 to 83]
  Stable Disease | 8 [2 to 21]
  Progressive Disease | 5 [1 to 17]

2. Secondary Outcome: Median Proportion Progression-free as Estimated by Kaplan-Meier Methods
Description: PFS was defined as time from trial enrollment to disease progression or death, whichever occurred first.
Time Frame: 5 years
Population: One subject lost to follow up and not included in analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane, Carboplatin, Bevacizumab
Number analyzed (Participants) | 40
months | 15 [10 to 25]

3. Secondary Outcome: To Evaluate Sequential Plasma Samples for Presence of Selected Angiogenic Markers
Time Frame: 18 months
Population: Analysis of samples was not performed, as there was inadequate funding to support the testing and analysis of the samples.
Arm/Group | Abraxane, Carboplatin, Bevacizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: to Determine if Apolipoprotein Alleles (Apo-E) Correlate With Treatment-related Neuropathy
Time Frame: 18 months
Population: Samples were collected, but analysis was not performed as there was inadequate funding to support the testing and analysis of samples.
Arm/Group | Abraxane, Carboplatin, Bevacizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: to Determine if SPARC Expression in Breast Tumors Predicts Progression-free Survival (PFS)
Time Frame: 18 months
Population: Study plan stipulated that tissue samples would not be assessed for quantitatively if no difference in SPARC expression was observed between tumor and non-tumor cells was observed qualitatively.
Arm/Group | Abraxane, Carboplatin, Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Abraxane, Carboplatin, Bevacizumab
Serious Adverse Events (participants affected / at risk) | 22/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane, Carboplatin, Bevacizumab (N=41)
Anemia (Blood and lymphatic system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Allergic reaction (Immune system disorders) | 1
Infections and infestations - Other, specify: (Infections and infestations) | 1 — Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Abdomen NOS
Vascular access complication (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 2
Nervous system disorders - Other, specify: Leptomeningeal Carcinomatosis (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: scalp discoloration (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane, Carboplatin, Bevacizumab (N=41)
Anemia (Blood and lymphatic system disorders) | 20
Blood and lymphatic system disorders - Other, specify: Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify: upper extremity lymphedema (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hemolysis (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 2
Cardiac disorders - Other, specify: Palpitations (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Ear and labyrinth disorders - Other, specify: Ringing in ears (Ear and labyrinth disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 6
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 6
Conjunctivitis (Eye disorders) | 1
Extraocular muscle paresis (Eye disorders) | 2
Eye disorders - Other, specify: vision changes (Eye disorders) | 3
Flashing lights (Eye disorders) | 1
Watering eyes (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 8
Anal fistula (Gastrointestinal disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Anal mucositis (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 25
Diarrhea (Gastrointestinal disorders) | 15
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 2
Esophageal pain (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify: dyspepsia (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 26
Oral pain (Gastrointestinal disorders) | 1
Rectal fistula (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Chills (General disorders) | 2
Edema face (General disorders) | 1
Edema limbs (General disorders) | 8
Edema trunk (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 34
Fever (General disorders) | 2
General disorders and administration site conditions - Other, specify: mouth sores (General disorders) | 7
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 16
Allergic reaction (Immune system disorders) | 3
Cytokine release syndrome (Immune system disorders) | 1
Anorectal infection (Infections and infestations) | 1
Bladder infection (Infections and infestations) | 1
Infections and infestations - Other, specify: (Infections and infestations) | 1 — Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Bladder (urinary)
Infections and infestations - Other, specify: (Infections and infestations) | 1 — Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Urinary tract NOS
Infections and infestations - Other, specify: URI/Sinusitis/laryngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Tooth infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Bruising (Injury, poisoning and procedural complications) | 1
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 1
INR increased (Investigations) | 1
Investigations - Other, specify: hypokalemia (Investigations) | 1
Neutrophil count decreased (Investigations) | 31
Platelet count decreased (Investigations) | 18
Weight gain (Investigations) | 2
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify: Cramping in Left Calf (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Ataxia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 12
Extrapyramidal disorder (Nervous system disorders) | 2
Glossopharyngeal nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 16
Memory impairment (Nervous system disorders) | 2
Nervous system disorders - Other, specify: Leptomeningeal Carcinomatosis (Nervous system disorders) | 2
Olfactory nerve disorder (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 23
Sinus pain (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 11
Insomnia (Psychiatric disorders) | 16
Personality change (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 2
Breast pain (Reproductive system and breast disorders) | 5
Ovulation pain (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 10
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 20
Dry skin (Skin and subcutaneous tissue disorders) | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Nail loss (Skin and subcutaneous tissue disorders) | 8
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10
Skin and subcutaneous tissue disorders - Other, specify: scalp discoloration (Skin and subcutaneous tissue disorders) | 11
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 3
Flushing (Vascular disorders) | 4
Hot flashes (Vascular disorders) | 14
Hypertension (Vascular disorders) | 5
Lymphedema (Vascular disorders) | 2
Vascular disorders - Other, specify: Nose bleed (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No